CLINICAL TRIAL: NCT00106964
Title: A Randomized, Open-Label Trial of Three Hepatitis B Vaccination Schemas in HIV-Positive Youth
Brief Title: Comparison of Three Hepatitis B Vaccination Regimens in HIV-Positive Youth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN 024
Record Dates: First submitted 2005-04-01; First posted 2005-04-04 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2016-02

CONDITIONS: HIV Infection; Hepatitis B
Keywords: Hepatitis B vaccines; HIV-infected adolescents; Hepatitis B infection (negative)
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Engerix-B; Hepatitis B Surface Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Standard dose (20 mcg) of Hepatitis B vaccine.
  Interventions: Biological: Engerix-B 20 mcg
- 2 (Active Comparator): 40 mcg of Hepatitis B vaccine
  Interventions: Biological: Engerix-B 40 mcg
- 3 (Active Comparator): 20 mgc of Twinrix
  Interventions: Biological: Twinrix 720 EIA HAV Ag plus 20 mcg HBsAg

INTERVENTIONS:
Biological: Engerix-B 20 mcg — A single dose of 1 mL (20 mcg/mL) will be administered in the deltoid muscle at Entry, Weeks 4 and 24.
  Arms: 1
Biological: Engerix-B 40 mcg — A single dose of 2 mL (20 mcg/mL) will be administered in the deltoid muscle at Entry, Week 4 and 24.
  Arms: 2
Biological: Twinrix 720 EIA HAV Ag plus 20 mcg HBsAg — Arm 3: 720 EIA HAV Ag, 20 mcg HBsAg/ml:
  A single dose of 1 mL will be administered in the deltoid muscle.
  Arms: 3

SUMMARY:
Hepatitis B is a contagious virus that can damage a person's liver. It can be prevented by vaccination, but for many HIV-positive people, the vaccines do not help them achieve adequate protection against this virus. In an attempt to improve response to vaccination and achieve protection from hepatitis B, this trial will compare the immune system response to 3 hepatitis B vaccine regimens in HIV-positive adolescents 12 through 24 years of age.

DETAILED DESCRIPTION:
Suboptimal response to hepatitis B vaccination in HIV+ adults and children has been well documented in the literature. Given the importance of preventing hepatitis B virus (HBV) co-infection in HIV+ youth and the poor response rates in this population, this study will attempt to improve the immediate and long-term sero-response rates by undertaking a randomized, open-label trial of three hepatitis B vaccination schemas, as follows:

1. standard adult dosing of HBV-only vaccine: Engerix-B 20 mcg at Entry, Week 4 and Week 24
2. increased adult dosing of HBV-only vaccine: Engerix-B 40 mcg at Entry, Week 4 and Week 24
3. standard adult dosing of combined HBV/hepatitis A virus (HAV) vaccine: Twinrix 720 enzyme immunoassay (EIA) HAV Ag plus 20 mcg HBsAg at Entry, Week 4 and Week 24.

This study will also describe the safety of administration of an increased dose of the hepatitis B vaccine in this population. In general, patients undergoing dialysis who have received the dosing regimen recommended for immunocompromised individuals have tolerated the vaccine series well.

Design: This is a stratified, block-randomized, open-label trial of three hepatitis B vaccination schemas in HIV-infected and HBV-uninfected youth. Once randomized, there will be a total of 6 study visits in a 72 week period. Vaccination will occur at Entry, Week 4 and Week 24. Primary sero-response will be evaluated at Week 28 and sustainability of response will be evaluated at Weeks 48 and 72 for those who achieve a primary antibody response of >= 10 IU/ml. Primary non-responders (antibody response of < 10 IU/ml) will be provided with a booster vaccine using the increased-dose Engerix-B vaccine at Week 48 and evaluated for responsiveness at Week 72.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV+
* Age 12 to < 25 years
* History of no or one hepatitis B vaccination
* Not pregnant.
* Females engaging in sexual intercourse must be willing to practice an approved method of birth control throughout the completion of the vaccine phase of the study.

Exclusion Criteria:

* History of > 1 hepatitis B vaccination
* Serologic evidence of past or present hepatitis B infection: anti-hepatitis B surface antigen (HBsAg), HBs-Ag or anti- hepatitis B core antigen (HBcAg)
* Previous allergic reaction to hepatitis A or B vaccinations or to yeast, thimerosal or aluminum.
* Active opportunistic infection or current treatment for known or suspected active serious bacterial infection at the pre-entry exam.

Presence of any known grade >= 3 clinical or laboratory toxicity at the time of pre-entry per toxicity tables.

* Anticipation of long-term corticosteroid therapy or within 3 months preceding study randomization. Use of non-steroidal, anti-inflammatory agents and inhaled or topical corticosteroids are allowed.
* Receipt of any restricted medicine listed in the protocol section 8.1.3 within 3 months preceding randomization.
* Receipt of immune globulin product or plasma product within 6 months preceding randomization
* Receipt of licensed blood product or transfusion or any licensed vaccine within 4 weeks preceding randomization.
* Known or suspected diseases of the immune system, other than HIV, or treatment for a malignancy within 3 months of randomization.
* Other serious, acute or chronic medical or surgical conditions must be approved by the protocol chair.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 371 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Flynn, MD, Study Chair — St. Jude Children's Research Hospital; Patricia Emmanuel, MD, Principal Investigator — University of South Florida, Peds. Div. of Infectious Disease; Diane M. Straub, MD, Principal Investigator — University of South Florida, Peds. Div. of Infectious Disease; Jorge Lujuan-Ziberman, MD, Principal Investigator — University of South Florida, Peds. Div. of Infectious Disease; Lawrence D'Angelo, MD, Principal Investigator — Children's National Medical Center, Div. of Aldol & Young Adult Medicine; Carleen Townsend-Akpan, CPNP, Principal Investigator — Children's National Medical Center, Div. of Aldol & Young Adult Medicine; Jaime Martinez, MD, Principal Investigator — John H. Stroger Jr. Hospital; Lisa Henry- Reid, MD, Principal Investigator — John H. Stroger Jr. Hospital; Irma Febo, MD, Principal Investigator — University Pediatric Hospital; LLeana Blasini, MD, Principal Investigator — University Pediatric Hospital; Donna Futterman, MD, Principal Investigator — Montefiore Medical Center; Marina Catallozzi, MD, Principal Investigator — Montifiore Medical Center; Linda Levin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Barbara Moscicki, MD, Principal Investigator — Univ. of California at San Franciso; Coco Auerswald, MD, Principal Investigator — Univ. of California at San Franciso; Sue Ellen Abdalian, MD, Principal Investigator — Tulane Medical Center; Ligia Peralta, MD, Principal Investigator — University of Maryland; Lawrence Friedman, MD, Principal Investigator — University of Miami; Ana Puga, MD, Principal Investigator — Children's Diagnostic & Treatment Center; Stephen Spector, MD, Principal Investigator — University of California, San Diego; Rolando M Viani, MD, Principal Investigator — University of California, San Diego
Locations (11):
- United States (4):
  - Childrens Hosp of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Children's Hosp Natinal Med Center, Washington D.C., District of Columbia
  - Tulane Med Center, New Orleans, Louisiana
- Brazil (5):
  - Federal University of Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto/USP, Ribeirão Preto, São Paulo
  - Instituto de Infectologia Emilio Ribas, São Paulo, São Paulo
  - Hospital dos Sevidores do Estado, Rio de Janeiro
  - Ippmg-Ufrj, Rio de Janeiro
- South Africa (2):
  - Tygerberg Hospital, Bellville, Cape Town
  - Harriet Shezi Childrens Clinic Chris Hani Baragwanth Hospital, Johannesburg, Gauteng

REFERENCES:
- [Result] Flynn PM, Cunningham CK, Rudy B, Wilson CM, Kapogiannis B, Worrell C, Bethel J, Monte D, Bojan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN). Hepatitis B vaccination in HIV-infected youth: a randomized trial of three regimens. J Acquir Immune Defic Syndr. 2011 Apr;56(4):325-32. doi: 10.1097/QAI.0b013e318203e9f2. PMID 21350366
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multi-site study. Accrual was open between April 2006 and January 2008. Participants were enrolled in the United States, South Africa, Brazil, and the Bahamas.
Pre-assignment Details: Subjects were randomized into one of three arms using blocks of six and stratified by absolute CD4 count (less than 500 and 500 cells/mL or greater) and previous hepatitis B virus (HBV) vaccination (0,1). The randomization was restricted so that the percentage of subjects with CD4 count < = 200 cells/mL would not exceed 15% of subjects on any arm.
Groups:
- 1: Engerix 20 mcg: Standard dose (20 mcg) of Hepatitis B vaccine. Dose #1 at Entry; Dose #2 at Week 4; Dose #3 at Week 24.
- 2: Engerix 40 mcg: 40 mcg of Hepatitis B vaccine. Dose #1 at Entry; Dose #2 at Week 4; Dose #3 at Week 24.
- 3: Twinrix 20 mcg: 20 mcg of Twinrix. Dose #1 at Entry; Dose #2 at Week 4; Dose #3 at Week 24.
Period: Overall Study
Arm/Group | 1: Engerix 20 mcg | 2: Engerix 40 mcg | 3: Twinrix 20 mcg
Started | 118 | 126 | 127
Completed | 105 (The number of those those who completed the vaccine series was 105.) | 111 (The number of those who completed the vaccine series was 111.) | 120 (The number of those who completed the vaccine series was 120.)
Not Completed | 13 | 15 | 7
Not completed — Lost to Follow-up | 8 | 6 | 2
Not completed — Pregnancy | 2 | 3 | 2
Not completed — Death | 1 | 1 | 0
Not completed — Incarceration | 0 | 1 | 0
Not completed — Site Funding Terminated | 0 | 1 | 1
Not completed — Failure to adhere | 2 | 0 | 0
Not completed — Did not meet eligibility criteria | 0 | 2 | 2
Not completed — Required disallowed medication | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Engerix 20 mcg | 2: Engerix 40 mcg | 3: Twinrix 20 mcg | Total
Number analyzed (Participants) | 118 | 126 | 127 | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.56 (3.42) | 20.96 (3.25) | 20.20 (3.50) | 20.57 (3.40)
Age, Customized [Number; unit: participants]
  12-13 years | 8 | 3 | 8 | 19
  14-15 years | 5 | 11 | 10 | 26
  16-19 years | 25 | 18 | 20 | 63
  >20 years | 80 | 94 | 89 | 263
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 74 | 80 | 227
  Male | 45 | 52 | 47 | 144
Region of Enrollment [Number; unit: participants]
  United States | 52 | 54 | 49 | 155
  South Africa | 4 | 6 | 13 | 23
  Brazil | 52 | 58 | 58 | 168
  Bahamas | 10 | 8 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Sero-response to Hepatitis B Surface Antigen
Description: The primary outcome, percentage positive sero-response, was compared between Arm 1 and each of the two alternative strategy arms (Arm 2 and Arm 3) and measured 4 weeks after the third vaccination at Week 28. Response is defined as greater than or equal to 10 IU/mL of serum being present; non-response is defined as less than 10 IU/mL.
Time Frame: Week 28
Population: Participants who completed a Week 28 visit with a Hepatitis B serology result were included in this analysis.
Measure: Number; unit: percentage of participants who resonded
Arm/Group | 1: Engerix 20 mcg | 2: Engerix 40 mcg | 3: Twinrix 20 mcg
Number analyzed (Participants) | 106 | 112 | 118
percentage of participants who resonded | 60 [0.00 to 0.00] | 73.2 [65 to 81.4] | 75.4 [67.7 to 83.2]
Statistical Analysis 1: Comparison: 1: Engerix 20 mcg vs 2: Engerix 40 mcg; Test type: Superiority or Other; p = 0.0440, Chi-squared
Statistical Analysis 2: Comparison: 1: Engerix 20 mcg vs 3: Twinrix 20 mcg; Test type: Superiority or Other; p = 0.0157, Chi-squared

2. Secondary Outcome: Safety of 3 Hepatitis B Vaccine Regimens in HIV+ Youth - ADVERSE EVENTS BY INTERVENTION ARM ON STUDY - POSSIBLY OR PROBABLY RELATED
Description: The number of adverse events (AE) was described by study arm. The proportion of subjects with clinical adverse events in Arms 1 and each of the two alternative strategy arms (Arm 2 and Arm 3) were compared to assess whether or not there is a difference in patients with any grade toxicity.
Time Frame: Baseline through Week 72
Population: All enrolled participants were included in this analysis of all AEs that were possibly or probably related to study drug. There were no AEs above Grade 3 considered to be possibly or probably related to study drug.
Measure: Number; unit: Events
Groups:
- 1: Engerix 20 mcg: Standard dose (20 mcg) of Hepatitis B vaccine. Number of participants with a Grade 1 event that was probably or possibly related to study drug as determined by the Site Investigator.
- 2: Engerix 40 mcg: Engerix 40 mcg vaccine. Number of participants with a Grade 1 event that was probably or possibly related to study drug as determined by the Site Investigator.
- 3: Twinrix 20 mcg: Twinrix 20 mcg vaccine. Number of participants with a Grade 1 event that was probably or possibly related to study drug as determined by the Site Investigator.
Arm/Group | 1: Engerix 20 mcg | 2: Engerix 40 mcg | 3: Twinrix 20 mcg
Number analyzed (Participants) | 118 | 126 | 127
Events
  Asthenia, Grade 1 | 0 | 0 | 1
  Arthralgia, Grade 3 | 1 | 0 | 0
  Headache, Grade 1 | 1 | 0 | 0
  Headache, Grade 2 | 2 | 0 | 0
  Somnolence, Grade 1 | 0 | 0 | 1
  Syncope Vasovagal, Grade 1 | 0 | 0 | 1

3. Secondary Outcome: Safety of 3 Hepatitis B Vaccine Regimens in HIV+ Youth - ADVERSE EVENTS BY INTERVENTION ARM ON STUDY - DEFINITELY RELATED
Description: The number of AEs was described by study arm. The proportion of subjects with clinical AEs in Arms 1 and each of the two alternative strategy arms (Arm 2 and Arm 3)were compared to assess whether or not there is a difference in subjects with any grade toxicity.
Time Frame: Baseline through Week 72
Population: All enrolled participants were included in this analysis of AEs that were definitely related to study drug. There were no AEs above Grade 2 considered to be definitely related to study drug.
Measure: Number; unit: event
Groups:
- 1: Engerix 20 mcg: Standard dose (20 mcg) of Hepatitis B vaccine. Number of participants with a Grade 1 event that was definitely related to study drug as determined by the Site Investigator.
- 2: Engerix 40 mcg: Engerix 40 mcg vaccine. Number of participants with a Grade 1 event that was definitely related to study drug as determined by the Site Investigator.
- 3: Twinrix 20 mcg: Twinrix 20 mcg vaccine. Number of participants with a Grade 1 event that was definitely related to study drug as determined by the Site Investigator.
Arm/Group | 1: Engerix 20 mcg | 2: Engerix 40 mcg | 3: Twinrix 20 mcg
Number analyzed (Participants) | 118 | 126 | 127
event
  Injection Site Pain, Grade 1 | 1 | 0 | 1
  Myalgia, Grade 2 | 1 | 0 | 1

4. Secondary Outcome: Safety of 3 Hepatitis B Vaccine Regimens in HIV+ Youth - ABNORMAL LABORATORY VALUES GRADE 2 OR ABOVE BY INTERVENTION ARM ON STUDY
Description: The number of adverse events and subjects with the events were described by study arm. The proportion of subjects with abnormal labs in Arms 1 and each of the two alternative strategy arms (Arm 2 and Arm 3) were compared to assess whether or not there is a difference in subjects with grade 3 or 4 toxicity. The laboratory events included are AEs classified as probably, possibly, or definitely related to study drug as classified by the Site Investigator.
Time Frame: Baseline through Week 72
Population: All enrolled participants were included in this analysis. The following no. of participants experienced at least one Grade 2 or higher abnormal labs by study arm.
Measure: Number; unit: Events
Units Other Than Participants: Events
Groups:
- 3: Twindrix 20 mcg: 20 mcg of Twinrix. Dose #1 at Entry; Dose #2 at Week 4; Dose #3 at Week 24.
Arm/Group | 1: Engerix 20 mcg | 2: Engerix 40 mcg | 3: Twindrix 20 mcg
Number analyzed (Participants) | 102 | 109 | 118
Number analyzed (Events) | 10 | 10 | 19
Events
  Absolute Neutrophil Count | 7 | 5 | 9
  Hemoglobin | 0 | 1 | 2
  Platelets | 0 | 2 | 1
  White Blood Cell count | 3 | 2 | 7

5. Secondary Outcome: Response Rates in HIV+ Youth Within Each Study Arm by Study Duration
Description: Within each arm, the duration of response in HIV-infected youth was analyzed for all subjects who were responders at 28 weeks. The possible values for response duration could be 20 weeks or less (responder at 28 weeks but not at 48 weeks), 20 to 44 weeks (responder at 28 and 48 weeks but not at 72 weeks), or greater than 44 weeks (responder at 28, 48, and 72 weeks). A response of greater than 20 weeks includes those who responded after 20 weeks, but whose exact response duration was unknown.
Time Frame: Entry through Week 72
Population: Population analyzed were those who had an antibody titer measured at Week 28.
Measure: Number; unit: percentage of participants who responded
Arm/Group | 1: Engerix 20 mcg | 2: Engerix 40 mcg | 3: Twinrix 20 mcg
Number analyzed (Participants) | 61 | 78 | 81
percentage of participants who responded
  <= 20 weeks | 27.87 | 19.23 | 22.22
  21 - 44 weeks | 3.28 | 7.69 | 11.11
  > 20 weeks | 4.92 | 12.82 | 3.70
  > 44 weeks | 63.93 | 60.26 | 62.96
Statistical Analysis 1: Comparison: 1: Engerix 20 mcg vs 2: Engerix 40 mcg; Test type: Superiority or Other; p = 0.5822, Regression, Cox; Hazard Ratio (HR) = 0.840
Statistical Analysis 2: Comparison: 1: Engerix 20 mcg vs 3: Twinrix 20 mcg; Test type: Superiority or Other; p = 0.8698, Regression, Cox; Hazard Ratio (HR) = 1.050

6. Secondary Outcome: Sero-Response to Hepatitis B Surface Antigen; Predictor: STUDY ARM
Description: Response rate associated with the participant's study arm, baseline CD4 count, and interaction term that reflects how subjects in Arm 2 responded differently depending on their CD4 count. Response is defined as greater than or equal to 10 IU/mL of serum being present; non-response is defined as less than 10 IU/mL.
Time Frame: Week 28
Population: All participants who had a Week 28 Hepatitis B serology result
Measure: Number; unit: percentage of participants who responded
Arm/Group | 2: Engerix 40 mcg | 1: Engerix 20 mcg | 3: Twinrix 20 mcg
Number analyzed (Participants) | 112 | 106 | 118
percentage of participants who responded | 73.2 [0.07 to 1.19] | 60 [1.00 to 1.00] | 75.4 [1.09 to 3.63]
Statistical Analysis 1: Comparison: 2: Engerix 40 mcg vs 1: Engerix 20 mcg; Test type: Superiority or Other; p = 0.0853, Regression, Logistic; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.07 to 1.19] — Adjusted odds ratio (OR) Odds ratio depends on CD4 count resulting from interaction. For example, OR=0.29 for CD4 count = 0; OR= 2.91 for CD4 count = 460 (median CD4 count for the evaluable study population)
Statistical Analysis 2: Comparison: 1: Engerix 20 mcg vs 3: Twinrix 20 mcg; Test type: Superiority or Other; p = 0.0244, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.09 to 3.63] — Adjusted odds ratio

ADVERSE EVENTS:
Time Frame: Data were collected over a three year time period.
Description: There were no Serious Adverse Events (SAE) to report
Groups:
- 3. Twinrix 20 mcg: 20 mcg of Twinrix. Dose #1 at Entry; Dose #2 at Week 4; Dose #3 at Week 24.
Arm/Group | 1: Engerix 20 mcg | 2: Engerix 40 mcg | 3. Twinrix 20 mcg
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/126 | 0/127
Other Adverse Events (participants affected / at risk) | 28/118 | 25/126 | 25/127
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Engerix 20 mcg (N=118) | 2: Engerix 40 mcg (N=126) | 3. Twinrix 20 mcg (N=127)
General Disorders and Administration Site Conditions (General disorders) | 14 (14) | 3 (3) | 7 (7)
Nervous System Disorders (Nervous system disorders) | 17 (17) | 14 (14) | 12 (12)
Gastrointestinal Disorders (Gastrointestinal disorders) | 4 (4) | 11 (11) | 1 (1)
Investigations (Investigations) | 12 (12) | 5 (5) | 9 (9)
Blood and lymphatic System Disorders (Blood and lymphatic system disorders) | 7 (7) | 5 (5) | 6 (6)
Infecions and Infestations (Infections and infestations) | 14 (14) | 12 (12) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by protocol team and AMLG.